CLINICAL TRIAL: NCT04186897
Title: Postendodontic Pain Following Occlusal Reduction in Mandibular Posterior Teeth: a Single-centre Randomized Controlled Trial
Brief Title: Occlusal Reduction Effect on Postendodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Suzan AW Amin, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ENDO-CU-2013-12-10
Record Dates: First submitted 2019-11-28; First posted 2019-12-05 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Symptomatic Irreversible Pulpitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occlusal reduction (Experimental): Occlusal contacts on the functional and non-functional cusps were reduced.
  Interventions: Procedure: Occlusal reduction
- No occlusal reduction (Sham Comparator): Occlusal surfaces kept intact. No actual occlusal reduction..
  Interventions: Procedure: Sham occlusal reduction

INTERVENTIONS:
Procedure: Occlusal reduction — Occlusal contacts on the functional and non-functional cusps were reduced.
  Arms: Occlusal reduction
Procedure: Sham occlusal reduction — The occlusal surface left intact. No actual occlusal reduction.
  Arms: No occlusal reduction

SUMMARY:
The aim of this study, thus, was to assess the effect of occlusal reduction on postendodontic pain after the first (post-instrumentation) and the second (post-obturation) visit in mandibular posterior teeth with symptomatic irreversible pulpitis and sensitivity to percussion treated in two visits.

DETAILED DESCRIPTION:
The purpose of this randomized clinical trial was to evaluate the effect of occlusal reduction on post-instrumentation and post-obturation pain in mandibular posterior teeth with symptomatic irreversible pulpitis and sensitivity to percussion treated in two visits. Three hundred and eight patients were included in this study. Inclusion criteria were posterior mandibular teeth having symptomatic irreversible pulpitis with sensitivity to percussion. Patients were randomized into two equal groups. In the intervention group, occlusal reduction was done, while, in the control group, the occlusal surfaces were left intact. Conventional endodontic treatment was performed in two visits using a rotary nickel-titanium system followed by the lateral-condensation obturation technique. Post-instrumentation pain was assessed after 6, 12, 24 and 48 hours following the first visit, and post-obturation pain after 6 and 12 hours following the second visit. Each patient received a pain diary to record their pain levels and rescue medication intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-65 years old.
* The diagnosis of symptomatic irreversible pulpitis with sensitivity to percussion.
* Posterior mandibular teeth.

Exclusion Criteria:

* Pregnant women.
* Patients who reported bruxism or clenching.
* Patients who took analgesics during the last 12 hours before treatment start.
* Teeth with no occlusal contact.
* Unrestorable teeth.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Post-instrumentation pain using a pain-measuring scale | 6 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured.
Post-instrumentation pain using a pain-measuring scale | 12 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured.
Post-instrumentation pain using a pain-measuring scale | 24 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured.
Post-instrumentation pain using a pain-measuring scale | 48 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured.
Post-obturation pain using a pain-measuring scale | 6 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured.
Post-obturation pain using a pain-measuring scale | 12 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured.

SECONDARY OUTCOMES:
Sham analgesic intake incidence | 7 days
  Sham medication intake incidence (Yes/No) taken as an initial rescue medication in case of postoperative pain.
Analgesic intake incidence | 7 days
  Analgesic intake incidence (Yes/No) as a rescue medication in case postoperative pain persisted after the sham analgesic intake.

CONTACTS AND LOCATIONS:
Overall Officials: Randa El Boghdadi, PhD, Study Chair — Cairo University

REFERENCES:
- [Background] Rosenberg PA, Babick PJ, Schertzer L, Leung A. The effect of occlusal reduction on pain after endodontic instrumentation. J Endod. 1998 Jul;24(7):492-6. doi: 10.1016/S0099-2399(98)80054-X. PMID 9693578
- [Background] Arslan H, Seckin F, Kurklu D, Karatas E, Yanikoglu N, Capar ID. The effect of various occlusal reduction levels on postoperative pain in teeth with symptomatic apical periodontitis using computerized analysis: a prospective, randomized, double-blind study. Clin Oral Investig. 2017 Apr;21(3):857-863. doi: 10.1007/s00784-016-1835-y. Epub 2016 Apr 30. PMID 27129585